CLINICAL TRIAL: NCT07197294
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for Neurodevelopmental Disorder With or Without Variable Brain Abnormalities (NEDBA) Due to MAPK8IP3 Mutation
Brief Title: Personalized Antisense Oligonucleotide for a Single Participant With MAPK8IP3 Neurodevelopmental Disorder With or Without Variable Brain Abnormalities (NEDBA)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV6360
Record Dates: First submitted 2025-07-23; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Neurodevelopmental Disorder With or Without Variable Brain Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-MAPK8-001

INTERVENTIONS:
Drug: nL-MAPK8-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with Neurodevelopmental Disorder with or without Brain Abnormalities (NEDBA) due to a heterozygous pathogenic missense mutation in MAPK8IP3

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with NEDBA due to a heterozygous pathogenic missense mutation in MAPK8IP3

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s)
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records
* Genetically confirmed neurodevelopmental disorder due to MAPK8IP3 mutation

Exclusion Criteria:

* Use of investigational medication within 5 half-lives of the drug at enrolment
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Ages: 5 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by the Gross Motor Function Measure-88 score.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by the Gross Motor Function Classification Scale (GMFCS) score.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by the Manual Ability Classification Scale (MACS) level.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by the Bayley Scales of Infant and Toddler Development 4th Edition (BSID-4) score.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by the Vineland Adaptive Behavior Scales - Third Edition (Vineland-3) score.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by distance, velocity, acceleration, movement shape, and entropy of movement captured on wrist and ankle accelerometers.

SECONDARY OUTCOMES:
Seizure Onset | Baseline to 24 months
  Change in presence of seizures from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by number of seizures recorded by EEG monitoring.
Seizure Onset | Baseline to 24 months
  Change in presence of seizures from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by changes in caregiver reported seizure tracker.
Respiratory Infections | Baseline to 24 months
  Change in frequency of treatment and hospitalizations for respiratory infection from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by changes in concomitant medications.
Respiratory Infections | Baseline to 24 months
  Change in frequency of treatment and hospitalizations for respiratory infection from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by frequence of adverse events.
Sleep Quality | Baseline to 24 months
  Change in sleep architecture from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured using an actigraphy device to monitor sleep duration.
Quality of Life | Baseline to 24 months
  Change in quality of life from baseline to 12- and 24-months post nL-MAPK8-001 administration as measured by Caregiver Global Impression of Change questionnaire (CaGI-C)
Safety and Tolerability | Baseline to 24 months
  Incidence and severity of treatment-emergent adverse events (AEs) from baseline to 12- and 24-months post nL-MAPK8-001 administration
Safety and Tolerability | Baseline to 24 months
  Changes from baseline to 12- and 24-months post nL-MAPK8-001 administration in physical examination (changes in appearance, skin, neck, ears, nose, throat, heart/lungs, abdomen, lymph nodes, and extremities compared to baseline)
Incidence of Treatment-Emergent Abnormalities in Neurological Exam [Safety and Tolerability] | Baseline to 24 months
  Changes from baseline to 12- and 24-months post nL-MAPK8-001 administration in neurological examination (changes in mental status, gait, cerebellar, cranial nerve, motor, reflex, and sensations compared to baseline as assessed by treating physician)
Incidence of Treatment Emergent Abnormalities in safety labs (CSF, chemistry, hematology, coagulation, urinalysis) [Safety and Tolerability] | Baseline to 24 months
  Emergent abnormalities in laboratory analyses (results outside of normal range for CSF, chemistry, hematology, coagulation, and urinalysis)

OTHER OUTCOMES:
Communication | Baseline to 24 months
  Change in communication skills from baseline to 6-, 12-, 18-, and 24-months post nL-MAPK8-002 administration as measured by Observer-Reported Communication Ability (ORCA)
Communication | Baseline to 24 months
  Change in communication skills from baseline to 12-, and 24-months post nL-MAPK8-002 administration as measured by Bayley Scales of Infant and Toddler Development 4th Edition (BSID-4)
Communication | Baseline to 24 months
  Change in communication skills from baseline to 12-, and 24-months post nL-MAPK8-002 administration as measured by Vineland Adaptive Behavior Scales - third Edition (Vineland-3)
Swallow function | Baseline to 24 months
  Change in swallow function from baseline to 12-, and 24-months post nL-MAPK8-002 administration as measured by a formal swallow study changes in oral and pharyngeal phases.
Swallow Function | Baseline to 24 months
  Change in swallow function from baseline to 12-, and 24-months post nL-MAPK8-002 administration as measured by Pediatric Functional Oral Intake Scale (pFOIS)
Swallow Function | Baseline to 24 months
  Change in swallow function from baseline to 12-, and 24-months post nL-MAPK8-002 administration as measured by Eating and Drinking Ability Classification System for individuals with CP (EDACS)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States